CLINICAL TRIAL: NCT00394264
Title: Manual Manipulative Therapy for Back Pain in Active Duty Military Personnel
Brief Title: How Does Manual Therapy Improve Low Back Pain for Soldiers?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: Samueli Institute for Information Biology (Other); Madigan Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1 EA-0000048; MILCAM-Madigan-Ft. Lewis
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2006-10-31 (Estimated); Status verified 2006-10

CONDITIONS: Low Back Pain
Keywords: low back pain; active duty military personnel; manual/manipulative therapy; osteopathic manipulative treatment; physical medicine
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy; Tocopherols

INTERVENTIONS:
Procedure: Soft Tissue
Procedure: Myofascial release
Procedure: Counterstrain
Procedure: Muscle energy
Procedure: Sacro-iliac articulation
Procedure: High-velocity, low amplitude

SUMMARY:
Musculoskeletal injuries including low back pain (LBP) are a major problem in military personnel. These injuries can result from training exercises, job duties, or recreational activities. However incurred, many of these injuries can result in limited duty in work or training, and can decrease military readiness.

The National Osteopathic Research Center (ORC) will examine the effectiveness of a specific set of Osteopathic Manipulative Treatment interventions referred to as Manual/Manipulative Therapy (M/MT) to reduce pain and improve functioning in young active duty military personnel.

The broad overall goal of this proposed research project is to determine the feasibility of conducting a larger clinical trial of Manual/Manipulative Therapy (M/MT) in restoring full performance in military personnel in the operational environment. A second goal is to estimate the treatment effect size of M/MT in this population.

The following two hypotheses will guide the data study:

* Hypothesis 1: Subjects receiving manual/manipulative therapy for low back pain will report less pain at two and four weeks than subjects in the control group.
* Hypothesis 2: Subjects receiving manual/manipulative therapy for low back pain will achieve greater functioning at two and four weeks than subjects in the control group.

DETAILED DESCRIPTION:
Musculoskeletal injuries are among the most common injuries in the military, and cause more soldiers to miss time from active duty than any other health condition.These injuries account for up to 20% of all clinic visits at Fort Sam Houston.Of these visits, up to 36% are back-related, resulting in lost duty time, lost training time, and a negative impact on military preparedness. It is of interest to the military to refine interventions that would effectively and efficiently treat back related injuries.

Osteopathic manipulative treatment (OMT) has been studied as a treatment for low back pain in both chronic and subacute presentations in a variety of situations. OMT has been found effective in decreasing medication use for back pain and improving pain and functioning.In a study on low back pain in the Navy, use of OMT significantly reduced time on light duty and sick-in-quarters time.

The National Osteopathic Research Center (ORC) proposes to examine the efficacy of a specific set of OMT interventions referred to in this proposal as Manual/Manipulative Therapy (M/MT) to reduce pain and improve functioning in young active duty military personnel.

The site for this study is the Madiagan Amry Medical Center at Fort Lewis, WA. We will sample the active duty personnel who present at the outpatient clinics at the Hospital with a complaint of low back pain. Osteopathic physicians will provide the M/MT.

Enough subjects will be enrolled and randomized in the study for a total of 100 to complete the trial in two groups: a treatment group receiving M/MT plus standard care (SC), and a control group receiving SC only. Standard care may include medications, back care education and exercise instructions, and/or limited duty. M/MT sessions will last approximately 15-20 minutes, and will be provided up to twice a week for up to four weeks. Standard care will be provided as needed.

Outcomes to be measured are pain and functionality. Pain measures include a Visual Analog Scale (VAS) and medication use. Function will be measured by the Back Pain Functional Scale (BPFS), Roland-Morris Questionnaire (RMQ), and time on modified duty. The VAS and duty status will be recorded at each visit. All other outcomes will be assessed at two and four weeks.

At the initial visit, we will also collect demographic data, medical history, information on quality of life using the SF-36, and subject treatment expectation. A subject satisfaction survey and a measure of overall improvement will be completed at two and four weeks.

The broad overall goal of this proposed research project is to determine the feasibility of conducting a larger clinical trial of Manual/Manipulative Therapy (M/MT) in restoring full performance in military personnel in the operational environment. A second goal is to estimate the treatment effect size of M/MT in this population.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military personnel
* Male and Female
* Age range 17-35
* Present with a new episode of low back pain (may be acute or new episode of chronic)

Exclusion Criteria:

* Pregnancy
* Any serious neurological, rheumatological, or orthopedic conditions such as spondylolysis, spondylolithesis,fracture, nerve impingement, tumors, or infections.
* Prior manipulative treatment for this episode LBP.
* Leg pain worse than back pain indicating possible radiculopathy.
* Clinical evidence of a leg length discrepancy greater than 13mm.
* Inability to give informed consent.
* Inability to follow course of care for four weeks.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2006-10; Study Completion 2007-10

PRIMARY OUTCOMES:
Pain
Functionality

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Stoll, D.O., Ph.D., Principal Investigator — Osteopathic Research Center University of North Texas Health Science Center; Douglas M Maurer, D.O., Principal Investigator — U.S. Army-Madigan Army Medical Center, Fort Lewis
Locations (1):
- Madigan Army Medical Center, Fort Lewis, Washington, United States